CLINICAL TRIAL: NCT04794361
Title: Management of Patients Suspected of COVID 19 With Ultra Low Dose Thoracic Scanner
Acronym: COVID-19 ULD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local 2020/JF1
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — pcr Covid-19 and viral load, inflammation marker (CRP)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The year 2020 was marked by the emergence of a new respiratory disease: COVID19 related to an infection with the coronavirus SARS-CoV-2 (name given by the WHO on February 11, 2020). Initially appearing in China, in the province of Hubei, this epidemic has rapidly spread to be declared a global pandemic on March 12, 2020 by the WHO.Given the current context of the COVID-19 epidemic, strict hygiene measures have been taken in scanning rooms with systematic bio-cleaning. Strategies have been modified as a matter of urgency, with changes in the practices of electro radiology manipulators who work in "isolation" to avoid contamination. The number of scanners has increased exponentially following the curve of the epidemic, making it more and more difficult to systematically check the images before the patient leaves the room. To ensure sufficient image quality for interpretation of all scans, a complementary acquisition in ULD, with very low exposure, was systematically added to the acquisition protocol. The standard acquisition in LD, associated with this acquisition in ULD remain well below the diagnostic reference thresholds dictated by the nuclear safety authority (NRD: 350 mGy.cm. In Nîmes: LD: 100 to 150 mGy.cm and ULD: < 15 mGy.cm). These two acquisitions allow us to avoid breathing and movement artifacts, etc., without having to have the patients return for a new scan in case of a bad acquisition. This avoids an overexposure of the staff to the risk of infection by the SARS-CoV-2 virus.

The main objective of this retrospective study is to evaluate the diagnostic performance of ULD vs. LD for the accurate diagnosis of COVID-19 pneumopathy which presents a particular ground glass pattern

Our study will demonstrate that the ULD scanner can be used in the search for COVID-19 pneumopathy and thus limit the exposure of patients to X-rays, especially since thoracic scans are often repeated.

DETAILED DESCRIPTION:
Main objective To evaluate the diagnostic performance of ULD vs. LD scanning for the diagnosis of COVID-19 lung disease.

Primary endpoint LD and ULD acquisitions will be anonymized and randomized in a read list. Double reading of scans in a randomized and blinded manner of the results of LD and ULD acquisitions of chest scans performed for suspected COVID-19 by 2 radiologists (one junior and one senior). Scans will be classified as non-COVID and COVID. The reference will be the LD scan. In case of discrepancy, a third senior radiologist will be asked and the decision will be made by consensus.

Secondary objectives

* Objective evaluation of image quality (signal, noise, contrast to noise ratio)
* Subjective evaluation of image quality and confidence in interpretation.
* Specific study of ground glass signal in ULD

Secondary evaluation criteria

* Measurement of signal and noise in the image using ROIs positioned in the lung, trachea, fat, which measure the average signal intensity and its standard deviation. These measurements will be performed on LD and ULD acquisitions at the same locations.
* Likert scale to subjectively assess image quality and confidence in the diagnosis.
* Specific measurement of signal and noise in the ground glass using ROI positioned within the ground glass that measures the average signal intensity and its standard deviation. This measurement will be performed on LD and ULD acquisitions at the same location.

Population concerned Patients of the Nîmes University Hospital who have had a prescription for a thoracic CT scan for suspected COVID-19 since March 5, 2020 (beginning of the COVID-19 protocol) and until April 5. Patients having had the LD and ULD acquisitions.

ELIGIBILITY:
Inclusion Criteria:

Patients having had the LD and ULD acquisitions

Exclusion Criteria:

* scanner not passed through the COVID circuit, no ULD acquisition performed

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from the Nîmes University Hospital who had a chest CT prescription for suspected COVID-19 since March 5, 2020 (start of the COVID-19 protocol) and until April 5
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
reading of LD and ULD acquisitions | day 1
  Diagnostic performance of ULD vs LD scanner for the diagnosis of COVID-19 pneumopathy

CONTACTS AND LOCATIONS:
Locations (1):
- Julien FRANDON, Nîmes, France